CLINICAL TRIAL: NCT07342335
Title: Understanding and Breaking Barriers to Research Access for Cancer Patients
Brief Title: Breaking Barriers to Research Access
Status: Recruiting | Type: Observational
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C1337; 321327 (Other: IRAS)
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Research Barriers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a need to improve accessibility to research and clinical trials within the NHS. Key groups are consistently under-represented in research: those from minority ethnic backgrounds, those with lower socio-economic status and those with impaired capacity. This leads to inequality of healthcare and an inequality of patient experience. Increasing access to research would not only broaden research opportunities and bridge gaps in health equality; diverse research representation means better understanding of disease mechanisms and greater generalisability of findings across the patient population. There are well described socio-economic issues across the region that we serve within Cheshire and Merseyside. This brings health challenges for patients. Clatterbridge Cancer Centre is a large networked cancer centre serving Cheshire and Merseyside using a hub model. Research is a core strategic theme; it is hugely important that we understand not only the areas and hotspots of cancer across the region, but also that our patients with those cancers can access a portfolio of research that serves a distinct patient need. Currently there is a lack of such triangulated information within the Trust, which may mean that patient need remains unmet. Therefore the research is designed to understand any barriers that patients may have in accessing research, in tandem with a demographic review and mapping of patient referral and access to the current trials portfolio. This will lead to a truly patient centred approach in accessing research.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years. No upper age limit
* A confirmed diagnosis of cancer
* Patient planned to or is receiving treatment at The Clatterbridge Cancer Centre NHS Foundation Trust
* Able to provide informed consent

Exclusion Criteria:

* Patients with severe co-morbidities considered by the screening team to interfere with the individual's ability to complete requirements of the study or to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A wide range of participants will be approached, in terms of age, location, disease site and demographics to give a fair reflection of the patient population
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Research Barrier Perception and Research Facilitator Perception | 12 Months
  The primary outcome measures for the questionnaire portion of the study are the overall scores on Research Barrier Perception (RBP: Questions 7 - 11) and Research Facilitator Perception (RFB: Questions 13 - 17). The predictor variable is deprivation, as measured by the IMD, 2019.

SECONDARY OUTCOMES:
Sub-scores of the Research Participation Questionnaire and are Treatment Perception Scores, Practical Consideration Scores Trust scores, Information scores and Impact scores, and their relationship with deprivation | 12 Months
  The secondary outcomes relate to the sub-scores of the Research Participation Questionnaire and are Treatment Perception Scores, Practical Consideration Scores Trust scores, Information scores and Impact scores, and their relationship with deprivation (IMD, 2019) will be assessed using a multivariate regression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Clatterbridge Cancer Centre, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No